CLINICAL TRIAL: NCT06658236
Title: Comparative Effects of Upper Extremity Proprioceptive Neuromuscular Facilitation and Chest Expansion Exercises on Thoracic Mobility in Children With Cerebral Palsy
Brief Title: Upper Extremity Proprioceptive Neuromuscular Facilitation and Chest Expansion Exercises in Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/Naima Khalid
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: chest cirtometry; Cerebral palsy; thoracic mobility; PNF of upper extremity; chest expansion; BPAT
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: It will be a randomized control trial in which non-probability convenient sampling will be used. Two groups will be formed in which participants will be randomly divided. Group A will receive upper Extremity proprioceptive neuromuscular facilitation. Group B will receive chest expansion exercises.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols, and possible efforts will be put to mask both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation Group (Experimental): Group A will perform PNF exercises using a yellow Thera-Band with a flexion-abduction-external rotation pattern, followed by extension-adduction-internal rotation, all with the elbow extended. The protocol includes three sets of 10 reps, with 60-second rest intervals conducted thrice a week for 12 weeks.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- Chest Expansion Exercise Group (Experimental): Group B was instructed to 1) breathe normally at rest; 2) perform upper extremity flexion, abduction, and external rotation with inhalation, followed by extension, adduction, and internal rotation with exhalation using a yellow Thera-Band. Subjects completed three sets of 10 repetitions with a 1-minute rest between sets thrice a week for 12 weeks.
  Interventions: Other: Chest Expansion Exercises

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — Group A will follow a PNF-based training protocol to enhance strength, flexibility, and coordination. The exercises include two main movement patterns: flexion-abduction-external rotation with the elbow extended and extension-adduction-internal rotation with the elbow extended. These patterns target the muscles around the shoulder and upper chest. A yellow Thera-Band adds light resistance, increasing muscle engagement. The protocol also employs the reversal of antagonists technique, alternating between opposing muscle groups for balanced development and improved coordination. Participants will complete three sets of ten repetitions per session, with a 60-second rest between sets. The program spans 12 weeks, with three weekly sessions, allowing for consistent progress and muscle recovery. This structured approach aims to improve functional mobility and the performance of activities involving similar movements, offering a comprehensive training strategy through PNF and resistance.
  Arms: Proprioceptive Neuromuscular Facilitation Group
Other: Chest Expansion Exercises — Group B participants followed a breathing-coordinated exercise protocol using a yellow Thera-Band to improve upper extremity function. The protocol began with subjects breathing generally at rest. They were then instructed to synchronize their movements with their breathing: performing upper extremity flexion, abduction, and external rotation during inhalation, followed by extension, adduction, and internal rotation during exhalation. This coordination between breathing and movement aimed to enhance muscle activation and control. Each session included three trials of ten repetitions for each exercise, with a 1-minute rest between trials. The protocol was conducted three times per week over 12 weeks. This approach was designed to promote strength, flexibility, and coordination in the upper body while integrating breath control, which may also support relaxation and better movement efficiency. The structured schedule ensures consistent practice and gradual improvement over the 12 weeks
  Arms: Chest Expansion Exercise Group

SUMMARY:
Thoracic mobility is the mobility of the thoracic spine, and the rib cage is often measured by the degree of thorax expansion during breathing. Thoracic mobility is affected by many reasons, such as breathing mechanics, muscle stiffness, a sedentary lifestyle, and poor posture. The risk of respiratory illness should be assessed in all individuals with Cerebral palsy. Poor mobility of the thoracic will lead to limited breathing capacity and difficulty in daily life activities. Increasing thoracic mobility enhances dynamic alignment and functional movement. Proprioceptive Neuromuscular Facilitation (PNF) of upper extremity and chest expansion exercise can improve thoracic mobility. In this method, a physiotherapeutic approach is used in muscle strengthening, lengthening, and endurance training. The study aims to analyze the effect of an upper limb training program based on PNF techniques and chest expansion exercises on the thoracic mobility of a cerebral palsy patient.

DETAILED DESCRIPTION:
The current study will be a randomized control trial; data will be collected from the Lahore Garrison Institute of Special Education. The study will include 14 patients who are equally divided into two groups and randomly allocated. Inclusion criteria for the study will be either gender of CP patients at Gross Motor Function Classification System level I to III, who had no orthopedic surgery in the last 6 months and have a diagnosis of CP by doctors. Patients with scoliosis and any acute or current respiratory infection or other respiratory conditions, such as asthma or influenza, will be excluded from the study. One experimental group will perform upper extremity PNF combined with elastic resistance bands; the other group will perform chest expansion exercises, which are upper extremity flexion, abduction, and external rotation exercises with an elastic band. The outcomes to be analyzed will be thoracic mobility. Data collection will be done before and after the intervention. Tools used for data collection will be Brompton BPAT breathing pattern assessment tool (BPAT) and chest cirtometry. Data will be analyzed through SPSS version 23.00.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System level of I to III.
* BPAT score ≥ 4.
* Either gender will be included

Exclusion Criteria:

* Recent chest infection.
* Children who are hospitalized
* Scoliosis
* No orthopedic surgery in last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The Brompton BPAT (Breathing Pattern Assessment Tool) | The BPAT is completed with the patient seated comfortably in a supported chair for at least 5 minutes, with data collection taking approximately 1 minute.
  The BPAT (Breathing Pattern Assessment Tool) is a structured method for recording data collected during a respiratory physiotherapy assessment. It evaluates several components: (i) chest and abdominal wall movement, (ii) the sound of inspiratory flow, (iii) the sound of expiratory flow, (iv) the pathway of inspiration and expiration, (v) signs of air hunger (such as yawning, sighing, and deeper breaths), (vi) respiratory rate (RR), and (vii) breathing rhythm. Each component is scored from 0 to 2, where 0 represents normal function, and 2 indicates severe Dysfunctional Breathing, resulting in a total score ranging from 0 to 14. The BPAT is completed with the patient seated comfortably in a supported chair for at least 5 minutes, with data collection taking approximately 1 minute. A BPAT score of 4 or higher has been validated as a threshold for diagnosing Breathing Pattern Disorder, with ROC analysis showing an AUC of 0.938 (0.885-0.991), 95% sensitivity, and 78% specificity.

SECONDARY OUTCOMES:
Measuring tape for measuring chest expansion | The test for measuring chest mobility using a non-stretch measuring tape typically takes about 5 to 10 minutes.
  Chest mobility will be assessed using a non-stretch measuring tape placed at the level of the xiphoid process, measuring both at rest and during maximal inhalation and exhalation. Interclass correlation coefficients for chest expansion measurements using the tape have been reported to range from 0.95 to 0.97, indicating high reliability.
Pediatric Sleep Questionnaire | The test for assessing pediatric Obstructive Sleep Apnea using the symptom scale typically takes about 10 to 15 minutes to complete. This duration includes the time required for the caregiver or parent to respond to the 22 symptom items and any necessary
  The scale consists of 22 symptom items that assess various aspects of pediatric Obstructive Sleep Apnea (OSA), including the frequency of snoring, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, and behaviours such as inattention or hyperactivity. It has demonstrated a sensitivity of 0.85 and a specificity of 0.87, indicating its effectiveness in identifying children at risk for OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Naima Khalid, MS*, Principal Investigator — Riphah International Univerisity
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No